CLINICAL TRIAL: NCT04618133
Title: Time-restricted Eating to Improve Body Fat Mass in Overweight and Obese Individuals with Morning Chronotype: a Randomized, Open-label, Multi-arm Trial
Brief Title: Time-restricted Eating in Morning Chronotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tinh-Hai Collet, MD (Other)
Responsible Party: Sponsor-Investigator, Tinh-Hai Collet, MD, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01439
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early time-restricted eating (Experimental): Duration: 12 weeks
  Interventions: Behavioral: Early time-restricted eating
- Late time-restricted eating (Experimental): Duration: 12 weeks
  Interventions: Behavioral: Late time-restricted eating
- Active control (Active Comparator): Duration: 12 weeks
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Early time-restricted eating — Participants will be advised to eat only during a selected window of 8 hours over the 24-hour cycle, i.e. from 6am to 2pm, with a 1-hour allowance according to their daily routine
  Other Names: Early TRE
  Arms: Early time-restricted eating
Behavioral: Late time-restricted eating — Participants will be advised to eat only during a selected window of 8 hours over the 24-hour cycle, i.e. from noon to 8pm, with a 1-hour allowance according to their daily routine
  Other Names: Late TRE
  Arms: Late time-restricted eating
Behavioral: Active control — Participants will be advised to eat a minimum of 3 meals over the 24-hour cycle, i.e. breakfast from 6am to 9am, lunch from 11am to 2pm, dinner from 6pm to 10pm. Snacks will be allowed between meals
  Arms: Active control

SUMMARY:
Overweight and obesity are highly prevalent conditions worldwide, despite active research of new interventions over decades. Current interventions include medications or bariatric surgery, but these approaches cannot be used in all patients and require clear indications and a close multidisciplinary management. Therefore most patients and physicians rely on lifestyle interventions, focusing on a balanced diet and physical exercise.

Recent studies have uncovered that energy metabolism is also regulated by circadian rhythms, which depend on spontaneous diurnal oscillations of the central clock, retinal sensing of ambient light, and daily feeding-fasting cycles. The chronotype has an influence on behavioral patterns, where some people describe that they are more alert in the morning or in the evening: The morning or evening chronotypes, respectively. However, in modern societies, many people are exposed to external cues in misalignment with their circadians clocks. The mismatch between the individual chronotype and the social/work life can lead to metabolic disorders.

Time-restricted eating (TRE), i.e. energy intake limited to certain windows of time without restricting calories, is an appealing approach because it proposes to realign the circadian clocks with external cues provided by the timing of food intake, thus leading to better metabolic outcomes.

The investigators speculate that the TRE intervention needs to be personalized to reach efficacy in a broader population. To tailor the TRE intervention to each individual and harmonize their eating patterns in accordance to their chronotype, the investigators plan to test early TRE vs. late TRE vs. active control in overweight and obese individuals with morning chronotype.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria

  * Men and premenopausal women
  * Age 25-50 years
  * BMI 25-34 kg/m2
  * Stable weight (maximum ± 2 kg of usual body weight) over the previous 3 months
  * Stable body fat mass (maximum ± 1 kg of body fat mass) during the run-in phase
  * Eating window ≥ 12 hours during the run-in phase
  * Morning chronotype
* Work-related criteria

  * Daytime work at least 3 days per week over the previous 1 month and planned during the study
* Study-related criteria

  * Able to give informed consent and follow the study procedures for the entire duration
  * Confident use of a smartphone and able to take regular pictures of food/drinks

Exclusion Criteria:

* Clinical criteria

  * Pregnant and breastfeeding women, plans for maternity during the study
  * On a diet, intermittent fasting, in a weight management program over the previous 3 months or planned during the study
  * Eating disorder(s) or prior bariatric surgery
  * Diabetes with hypoglycemic drug(s)
  * Major illness/fever over the previous 1 month
  * Active major cardiovascular, respiratory, liver, gastrointestinal, renal, neurological or endocrine disorders
  * Coagulation disorder, on anticoagulant drug, skin disorder affecting wound healing
  * Active cancer and/or oncologic treatment over the previous 12 months
  * Major sleep disorder (including untreated sleep apnea syndrome), major mental illness
  * Consumption of > 7 standard units of alcohol per week for women and > 14 standard units of alcohol per week for men
* Work and time-related criteria

  * Shift work, such as evening shifts or night shifts, over the previous 1 month or planned during the study
  * Travel/trip to a different time zone (≥ 2-hour time difference) over the previous 1 month or planned during the study
* Study-related criteria and other interventions

  * Enrolled in another interventional clinical trial (medication, medical device) over the previous 1 month and planned during the study
  * Regular medications over the previous 1 month that could affect the study endpoints (e.g. centrally acting, medications affecting gut absorption, transit or weight, hypoglycemic drug, hormonal treatment...)

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Change in body fat mass | From randomization visit to close-out visit (12 weeks)
  As measured by dual-energy x-rax absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in physical activity | From randomization visit to close-out visit (12 weeks)
  As measured by actigraphy
Change in sleep/wake cycles | From randomization visit to close-out visit (12 weeks)
  As measured by actigraphy
Change in ambient light | From randomization visit to close-out visit (12 weeks)
  As measured by actigraphy
Change in sleep quality | From randomization visit to close-out visit (12 weeks)
  As measured by the Pittsburgh Sleep Quality Index (scale 0-21, 0 indicating no sleeping difficulty, 21 indicating severe sleeping difficulties)
Change in eating duration | From randomization visit to close-out visit (12 weeks)
  Duration from the first to last caloric intake over 24-hour cycle
Change in calorie intake over the 24-hour cycle | From randomization visit to close-out visit (12 weeks)
  Assessed by a 24-hour food recall
Change in weight | From randomization visit to close-out visit (12 weeks)
  Body weight (kg)
Change in waist circumference | From randomization visit to close-out visit (12 weeks)
  Waist circumference (cm) assessed with a measuring tape
Change in hip circumference | From randomization visit to close-out visit (12 weeks)
  Hip circumference (cm) assessed with a measuring tape
Change in systolic and diastolic blood pressure | From randomization visit to close-out visit (12 weeks)
  As measured with an arm cuff in the sitting position
Change in fasting glucose | From randomization visit to close-out visit (12 weeks)
  As measured in clinical chemistry
Change in lipid profile (concentration of total cholesterol, LDL cholesterol, triglycerides, HDL cholesterol) | From randomization visit to close-out visit (12 weeks)
  As measured by clinical chemistry
Change in body fat mass | From randomization visit to close-out visit (12 weeks)
  As measured by bioelectrical impedance analysis (BIA)
Change in lean body mass | From randomization visit to close-out visit (12 weeks)
  As measured by dual-energy x-rax absorptiometry (DXA)
Change in fat-free mass | From randomization visit to close-out visit (12 weeks)
  As measured by bioelectrical impedance analysis (BIA)
Change in resting energy expenditure | From randomization visit to close-out visit (12 weeks)
  As measured by indirect calorimetry
Change in glucose excursion | From randomization visit to close-out visit (12 weeks)
  As measured by continuous glucose monitoring
Incidence of adverse events in response to the randomized intervention | From randomization visit to close-out visit (12 weeks)
  Adverse events graded after the Common Terminology Criteria for Adverse Events version 5.0

OTHER OUTCOMES:
Change in in vitro circadian parameters (amplitude and magnitude) | From randomization visit to close-out visit (12 weeks)
  As measured in cultured skin fibroblasts (in a subset of the study population)
Change in metabolomic parameters | From randomization visit to close-out visit (12 weeks)
  As measured by high-throughput mass spectrometry metabolomics
Change in lipid metabolism | From randomization visit to close-out visit (12 weeks)
  As measured by high-throughput mass spectrometry lipidomics
Change in blood hormonal profile | From randomization visit to close-out visit (12 weeks)
  Cortisol, insulin, thyroid-stimulating hormone

CONTACTS AND LOCATIONS:
Overall Officials: Tinh-Hai Collet, MD, Principal Investigator — Geneva University Hospitals, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland